CLINICAL TRIAL: NCT02982603
Title: The Efficacy and Safety of Qinggongshoutao Bolus for aMnestic Mild Cognitive Impairment: A 52- Week Randomized, Double-blind, Controlled,Three Arms, Multi-center Study
Brief Title: Efficacy and Safety of Qinggongshoutao Bolus in aMnestic Mild Cognitive Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Clinical Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z12020286
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2015-05

CONDITIONS: Mild Cognitive Impairment; Herbal Medicine Allergy
MeSH Terms: conditions — Cognitive Dysfunction | interventions — ginaton; Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Qinggongshoutao Bolus (Experimental): Qinggongshoutao bolus and placebo identified to Ginkgo Biloba Extract 761 .Qinggongshoutao bolus 70 pills every time (7g), 2 times per day and placebo identified to Ginkgo Biloba Extract 761, 2 pills per time, 2 times per day for 48 weeks.
  Interventions: Drug: Qinggongshoutao Bolus
- Ginkgo Biloba Extract 761 (Active Comparator): Ginkgo Biloba Extract 761 and placebo identified to Qinggongshoutao bolus.The subjects will take Ginkgo Biloba Extract 761 2 times per day, 2 pills per time(80mg) ,and identified to Qinggongshoutao bolus 70 pills every time, 2 times per day for 48 weeks.
  Interventions: Drug: Ginkgo Biloba Extract 761
- Placebos (Placebo Comparator): Placebo identified to Qinggongshoutao bolus and placebo identified to Ginkgo Biloba Extract 761.Placebo identified to Qinggongshoutao bolus 70 pills every time, 2 times per day and placebo identified to Ginkgo Biloba Extract 761, 2 pills per time, 2 times per day for 48 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Qinggongshoutao Bolus — Qinggongshoutao bolus and placebo identified to Ginkgo Biloba Extract 761
  Other Names: Ginkgo biloba also named Egb761 or Ginaton
  Arms: Qinggongshoutao Bolus
Drug: Ginkgo Biloba Extract 761 — Placebo identified to Qinggongshoutao bolus and Ginkgo Biloba Extract 761
  Other Names: Ginkgo biloba also named Egb761 or Ginaton
  Arms: Ginkgo Biloba Extract 761
Drug: Placebos — Placebo identified to Qinggongshoutao Bolus and placebo identified to Ginkgo biloba
  Arms: Placebos

SUMMARY:
This study is a 52-weeks, multicenter, randomized, double-blind, double- placebo, parallel controlled phase VI trial being carried out in 20 centers around China. The study population includes amnestic mild cognitive impairment patients (planned a total of 360) aged 55-85 in both gender. Participants will be randomly allocated to Qinggongshoutao bolus (7g per time,2 times per day) and placebo identified to Ginkgo biloba (Ginaton), Ginkgo biloba (Ginaton) (80mg per time, 2 times per day) and placebo identified to Qinggongshoutao bolus, or placebo identified to Qinggongshoutao bolus and placebo identified to Ginkgo biloba (Ginaton) for a 52-weeks double-blind treatment period. The primary outcome measure is change from baseline in the Alzheimer's Disease Assessment Scale- Cognition Subscale (ADAS-cog) and rate of conversion to dementia. The secondary outcomes are changes from baseline in the Mini-Mental State Examination(MMSE), Delayed Story Recall(DSR), Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24). Safety is being assessed by observing side effects and adverse reaction during the entire treatment period. Statistical analysis will be conducted according to per-protocol population and intend-to-treat population and the safety will be analyzed in safety set.

ELIGIBILITY:
Inclusion Criteria:

1. cognitive complaints from the patients or their families;
2. objective evidence for memory impairment, delayed story recall test(DSR)<12.6(age50-64 less than15.5,65-74less than 12.5,older 75 less than10);
3. normal general cognitive function, with Mini-Mental State Examination (MMSE) score of between 24 and 30 (including 30);
4. preservation of activities of daily living, with Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24) score between 38 and 52;
5. cognitive disorders as evidenced by clinical evaluation, with clinical dementia rating scale=0.5,memory domain = 0.5;
6. absence of dementia, not sufficiently impaired cognitively and functionally to meet DSM-IV criteria,
7. enough vision and hearing to accomplishment neuropsychological test;
8. capability to read words and write simple sentence;
9. capability and willingness to give informed consent and to comply with the study procedures.

Exclusion Criteria:

1. non amnestic Mild cognitive impairment;
2. meeting the diagnostic criteria for dementia;
3. cognitive impairment resulting from conditions such as acute cerebral trauma, cerebral damage due to a lack of oxygen, epilepsy vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation, or a brain tumor ,or drug abuse or alcohol abuse
4. having significant psychiatric disease, depression, the Hamilton depression scale >12; CT or MRI scan showed central nervous system infections Infarction or focal lesions within 12 months，the Hachinski Ischemic Scale (HIS)>4;
5. combined following disease: diabetes; poor controlled hypertension or severe arrhythmias; or suffered from heart infarction within 3 months; severe asthma or COPD; severe indigestion; gastrointestinal tract obstruction; gastroduodenal ulcer;
6. used cholinesterase inhibitors or memantine within 1 month;
7. history of hypersensitivity to the treatment drugs;
8. concomitant drugs with the potential to interfere with cognition;
9. administration of other investigational drugs; severe impairment of the functions of the kidney or liver;
10. vegetarians or contraindications for animal innards.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of double-blind treatment of Alzheimer Disease Assessment Scale-cognitive subscale | week 0, week 4, week 12, week 24 ,week 36 , week 48 and week 52.
Change from baseline to end of double-blind treatment of rate of conversion to dementia | week 0, week 4, week 12, week 24 ,week 36 , week 48 and week 52.

SECONDARY OUTCOMES:
Mini-Mental State Examination(MMSE) | week 0, week 4, week 12, week 24 ,week 36 , week 48 and week 52.
Change from baseline to end of double-blind treatment of Delayed Story Recall test (DSR) | week 0, week 4, week 12, week 24 ,week 36 , week 48 and week 52.
Change from baseline to end of double-blind treatment of Alzheimer's Disease Cooperative Study/Activities of Daily Living scale adapted for MCI patients (ADCS/MCI/ADL24) | week 0, week 4, week 12, week 24 ,week 36 , week 48 and week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, M.D,PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital ,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No